CLINICAL TRIAL: NCT03341520
Title: Therapy of Nodal Follicular Lymphoma (WHO Grade 1/2) in Clinical Stage I/II Using Response Adapted Involved Site Radiotherapy in Combination With Gazyvaro
Brief Title: Gazyvaro and Low Dose Radiotherapy in Early Stage Follicular Lymphoma
Acronym: GAZAI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Principal investigator, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002059-89
Record Dates: First submitted 2017-11-06; First posted 2017-11-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Stage II Grade 1 Follicular Lymphoma; Stage II Grade 2 Follicular Lymphoma; Stage I Follicular Lymphoma Grade 1; Stage II Follicular Lymphoma Grade 2
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obinutuzumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Open, non-controlled, national multi-center phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- interventional arm (Experimental): Obinutuzumab Injection [Gazyva] 1000mg flat i.v. on week 1, 2, 3, 4, 8, 12, 16; Low dose radiation Therapy (LDRT) involved site 2 x 2 Gy in week 9
  Interventions: Drug: Obinutuzumab Injection [Gazyva]; Radiation: Low dose radiation Therapy (LDRT)

INTERVENTIONS:
Drug: Obinutuzumab Injection [Gazyva] — 7x 1000mg flat dose
  Other Names: Gazyvaro
Radiation: Low dose radiation Therapy (LDRT) — 2 x 2 Gy

SUMMARY:
Combined modality approach using Obitunuzumab and involved site low dose irradiation in early stage nodal follicular lymphoma. Radiation dose will be adapted for low-responders.

Primary Objective:

Evaluation of the rate of metabolic CR after low-dose involved site radiotherapy in combination with Gazyvaro (Obinutuzumab) in early stage nodal follicular lymphoma in order to avoid conventional full dose IF radiotherapy.

Secondary Objective:

Efficacy and safety of a response adapted radiation dose treatment schedule.

DETAILED DESCRIPTION:
Extended field or total nodal irradiation had been the gold standard for early stage follicular lymphoma for a long time in Germany. An involved field (IF) irradiation has been favored due to the toxicity of large field irradiation in other countries (e.g. USA). However, smaller irradiation fields have been accompanied with an increased risk of recurrence. A combination of involved field irradiation with the anti-CD20 antibody Rituximab (MIR trial) has led to similar efficacy results compared to the large field irradiation but with markedly reduced side effects.

Haas et al. showed in a prospective trial, that a low dose radiation therapy (LDRT) can lead to a complete remission in up to 60% in follicular lymphoma. This is presumed to result from immune modulatory effects induced by LDRT. The effectiveness of LDRT could also be demonstrated in another prospective, randomized British trial (FORT trial: 2 x2 Gy vs. 12 x 2 Gy) with a CR rate of 40% after 2 x 2 Gy (60% after 12 x 2 Gy). Currently, it is unknown, which patients need a higher radiation dose and which not.

A metabolic complete remission (CR) is an important prognostic marker for progression-free survival. According to the results of the PRIMA trial, CR is a very strong predictive parameter if the CR is established using FDG-PET.

In the present GAZAI trial, patients with early stage nodular follicular lymphoma will be treated in a combined approach of immunotherapy with an anti-CD20 antibody and small field (involved site) irradiation as in the MIR trial. In GAZAI, the fully humanized anti-CD20 antibody Obinutuzumab (GAZYVARO) will be used, which showed a high efficacy in combination with bendamustin in patients with follicular lymphoma refractory to Rituximab (GADOLIN trial). In addition, the radiation dose will be limited to 2 x2 Gy in responding patients. A dose build-up to a total of 40 Gy (dose in the MIR trial) will be performed in case of failure to achieve a complete CR based on a FDG-PET in week 18.

Primary endpoint of the trial is the rate of CR (based on FDG-PET/CT) after Obinutuzumab and 2x2 Gy IS radiotherapy in week 18. Secondary endpoints are the morphological CR rate in week 7, week 18 and month 6, the PFS, the toxicity, the recurrence rate, the recurrence pattern, overall survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Centrally reviewed CD20-positive follicular lymphoma grade 1/2 based on WHO classification (2016)
* Untreated (radiation-, chemo- or immunotherapy) nodal lymphoma (including involvement of Waldeyer´s ring)
* Age: ≥18 years
* ECOG: 0-2
* Stage: clinical stage I or II (Ann Arbor classification)
* Risk profile: Largest diameter of the lymphoma * 7 cm (sectional images)
* Written informed consent and willingness to cooperate during the course of the trial
* Adequate hematologic function (unless abnormalities are related to NHL), defined as follows: Hemoglobin ≥ 9.0 g/dL; absolute neutrophil count ≥ 1.5 × 109/L, Platelet count ≥ 75 × 109/L
* Capability to understand the intention and the consequences of the clinical trial
* Adequate contraception for men and women of child-bearing age during therapy and 18 months thereafter
* Patients with non-active hepatitis B infection (HBsAg neg/HBcAB pos/HBV DNA neg) under 1-year require prophylactic anti-viral therapy (e.g. Entecavir®) possible (see also 5.6. Prior and Concomitant Disease)

Exclusion Criteria:

* Extra nodal manifestation
* Secondary cancer in the patient's medical history (exclusion: basalioma, spinalioma, melanoma in situ, bladder cancer T1a, non-metastasized solid tumor in constant remission, which was diagnosed >3 years ago
* Concomitant diseases: congenital or acquired immune-deficiency syndromes, active infections including viral hepatitis (serology positive for HBsAg or HBcAb in combination positive HBV DNA), uncontrolled concomitant diseases including significant cardiovascular or pulmonary disease (see also 5.6. Prior and Concomitant Disease)
* Severe psychiatric disease
* Pregnancy / lactation
* Known hypersensitivity against Gazyvaro (Obinutuzumab) or drugs with similar chemical structure or any other additive of the pharmaceutical formula of the study drug
* Participation in another interventional trial or follow-up period of a competing trial which can influence the results of this current trial
* Creatinine > 1.5 times the upper limit of normal (ULN) (unless creatinine clearance normal), or calculated creatinine clearance < 40 mL/min
* AST or ALT > 2.5 × ULN
* Total bilirubin ≥ 1.5 × ULN
* INR > 1.5 × ULN
* PTT or aPTT > 1.5 × the ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Rate of metabolic complete remission (CR) | week 18
  rate of metabolic complete remission (CR) after low-dose involved site radiotherapy in combination with Obinutuzumab in patients with initially remaining PET positive lymphoma

SECONDARY OUTCOMES:
Rate of morphologic complete remission (CR) | week 7, week 18, month 6
  rate of morphologic complete remission (CR) after low-dose involved site radiotherapy in combination with Obinutuzumab in patients with initially remaining lymphoma
Progression free survival (PFS) | 2 years
  PFS of all patients
Toxicity | Start until month 30
  Common Toxicity Criteria (CTC) Toxicity
Overall survival (OS) | 2 years
  OS of all patients
Relapse rate | start until month 30
  Relapse rate of all patients
Quality of life (QoL) EORTC QLQ-C30 | Initially, week 18, month 12, month 24
  QoL according EORTC QLQ-C30
Minimal residual disease (MRD) response | initially, week 18, month 6, month 12, month 18, month 24
  Minimal residual disease
Relapse pattern | start until month 30
  Relapse pattern (e.g. out-field or in-field) of all relapses
Quality of life (QoL) FACT-Lymph25 | Initially, week 18, month 12, month 24
  QoL according FACT-Lymph25 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, MD, Study Chair — Radiation Therapy, University Hospital of Heidelberg ,Germany
Locations (12):
- Germany (12):
  - University of Tuebingen, Tübingen, Baden-Wurttemberg
  - Vivantes Klinikum, Berlin
  - University of Cologne, Cologne
  - University of Essen, Essen
  - University of Frankfurt, Frankfurt
  - University of Heidelberg, Heidelberg
  - Klinikum Kempten, Kempten
  - Site Marburg, Marburg
  - LMU, Munich
  - TU, Munich
  - University of Muenster, Münster
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mac Manus MP, Hoppe RT. Is radiotherapy curative for stage I and II low-grade follicular lymphoma? Results of a long-term follow-up study of patients treated at Stanford University. J Clin Oncol. 1996 Apr;14(4):1282-90. doi: 10.1200/JCO.1996.14.4.1282. PMID 8648385
- [Background] Haas RL, Poortmans P, de Jong D, Aleman BM, Dewit LG, Verheij M, Hart AA, van Oers MH, van der Hulst M, Baars JW, Bartelink H. High response rates and lasting remissions after low-dose involved field radiotherapy in indolent lymphomas. J Clin Oncol. 2003 Jul 1;21(13):2474-80. doi: 10.1200/JCO.2003.09.542. PMID 12829665
- [Background] Hoskin PJ, Kirkwood AA, Popova B, Smith P, Robinson M, Gallop-Evans E, Coltart S, Illidge T, Madhavan K, Brammer C, Diez P, Jack A, Syndikus I. 4 Gy versus 24 Gy radiotherapy for patients with indolent lymphoma (FORT): a randomised phase 3 non-inferiority trial. Lancet Oncol. 2014 Apr;15(4):457-63. doi: 10.1016/S1470-2045(14)70036-1. Epub 2014 Feb 24. PMID 24572077
- [Background] Trotman J, Fournier M, Lamy T, Seymour JF, Sonet A, Janikova A, Shpilberg O, Gyan E, Tilly H, Estell J, Forsyth C, Decaudin D, Fabiani B, Gabarre J, Salles B, Van Den Neste E, Canioni D, Garin E, Fulham M, Vander Borght T, Salles G. Positron emission tomography-computed tomography (PET-CT) after induction therapy is highly predictive of patient outcome in follicular lymphoma: analysis of PET-CT in a subset of PRIMA trial participants. J Clin Oncol. 2011 Aug 10;29(23):3194-200. doi: 10.1200/JCO.2011.35.0736. Epub 2011 Jul 11. PMID 21747087
- [Background] Sehn LH, Chua N, Mayer J, Dueck G, Trneny M, Bouabdallah K, Fowler N, Delwail V, Press O, Salles G, Gribben J, Lennard A, Lugtenburg PJ, Dimier N, Wassner-Fritsch E, Fingerle-Rowson G, Cheson BD. Obinutuzumab plus bendamustine versus bendamustine monotherapy in patients with rituximab-refractory indolent non-Hodgkin lymphoma (GADOLIN): a randomised, controlled, open-label, multicentre, phase 3 trial. Lancet Oncol. 2016 Aug;17(8):1081-1093. doi: 10.1016/S1470-2045(16)30097-3. Epub 2016 Jun 23. PMID 27345636
- [Derived] Konig L, Dreyling M, Durig J, Engelhard M, Hohloch K, Viardot A, Witzens-Harig M, Kieser M, Klapper W, Pott C, Herfarth K. Therapy of nodal Follicular Lymphoma (WHO grade 1/2) in clinical stage I/II using response adapted Involved Site Radiotherapy in combination with Obinutuzumab (Gazyvaro) - GAZAI Trial (GAZyvaro and response adapted Involved-site Radiotherapy): a study protocol for a single-arm, non-randomized, open, national, multi-center phase II trial. Trials. 2019 Aug 30;20(1):544. doi: 10.1186/s13063-019-3614-y. PMID 31470902

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT03341520/Prot_SAP_000.pdf